CLINICAL TRIAL: NCT05008991
Title: Assessment of Lung Functions in Menopausal Obese Women After COVID 19 Recovery
Brief Title: Lung Functions in Menopausal Obese Women After COVID 19 Recovery
Status: Completed | Type: Observational
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Hend Reda Sakr, Lecturer at Department of Physical Therapy for Woman's Health, Badr University
Other Study IDs: Hend 2
Record Dates: First submitted 2021-08-16; First posted 2021-08-17 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Lung Function Decreased; Obesity; Menopause; Covid19
Keywords: Lung funnctions; Menopause; Obesity; Covid19
MeSH Terms: conditions — Respiratory Insufficiency; Obesity; COVID-19 | interventions — Spirometry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: The study group will consist of (20) obese menopausal women whom are recently recovered from mild-moderate COVID-19 after one month.
  Interventions: Device: Spirometry
- Control group: The control group will consist of (20) obese menopausal women; whom are not be affected by COVID-19.
  Interventions: Device: Spirometry

INTERVENTIONS:
Device: Spirometry — Spirometry assesses the integrated mechanical function of the lung, chest wall, respiratory muscles, and airways by measuring the total volume of air exhaled from a full lung (total lung capacity [TLC]) to maximal expiration (residual volume [RV]). This volume, the forced vital capacity (FVC) and the forced expiratory volume in the first second of the forceful exhalation (FEV1), should be repeatable to within 0.15 L upon repeat efforts in the same measurement unless the largest value for either parameter is less than 1 L. In this case, the expected repeatability is to within 0.1 L of the largest value.

SUMMARY:
The COVID-19 pandemic has presented considerable challenges to global health services and dictates almost every aspect of medical practice and policy. The menopausal transition may have significant consequences for respiratory health as COVID 19 symptoms subsides, lung function testing should be done to assess the consequences of this virus on lung health especially in menopausal woman.

DETAILED DESCRIPTION:
The study group will consist of (40) obese menopausal women whom were recently recovered from mild-moderate COVID 19 for one month. The control group will consist of (40) obese menopausal women; whom will not affected by COVID 19. Using incentive spirometer, we will measure forced vital capacity FVC, forced expiratory volume FEV, Tiffano index TI and peak expiratory force PEF in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Participants recovered from mild to moderated signs and symptoms of COVID- 19 after one month.
* Ability to perform pulmonary function tests correctly.
* COVID-19 was diagnosed by positive polymerase chain reaction (PCR) testing on nasopharyngeal swab, oxygen saturation was ranged between 92-96% during illness period.
* CT chest shows ground glass opacity.
* Their D-dimer was less than 0.5 μg/ml.
* Two successive negative PCR were before included in study.
* Participants were in home isolation during illness period.

Exclusion Criteria:

* Chronic respiratory disease.
* Chronic heart disease.
* Diabetes mellitus.
* Smoking.
* Centralized isolation.
* Severe COVID-19.

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female menopausal women only.
Study Population: all women will be aged from 45 to 55 years old in menopause, their BMI will be from 30 to 34.9 kg/m2.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in the first second (FEV1) | FEV1 will be measured after 1 month post COVID19 recovery.
  is a measurement of your ability to expel air from your lungs. More specifically, and as its name suggests, it is the amount that is exhaled in the first second of purposefully trying to breathe out as much air as possible.
forced vital capacity (FVC) | FVC will be measured after 1 month post COVID19 recovery.
  is the total amount of air exhaled during the FEV test.
FEV1/FVC ratio | FEV1/FVC ratio will be measured after 1 month post COVID19 recovery.
  The FEV1/FVC ratio, also called Tiffeneau-Pinelli index, is a calculated ratio used in the diagnosis of obstructive and restrictive lung disease. It represents the proportion of a person's vital capacity that they are able to expire in the first second of forced expiration to the full, forced vital capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Mariam El Ebrashy, PhD, Principal Investigator — Badr University in Cairo
Locations (1):
- Faculty of Physical Therapy, Badr University, Cairo, New Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided